CLINICAL TRIAL: NCT03577951
Title: Comparing the Two Ways of Creating a High Position and Low Position Operating Space in Endoscopic Thyroid Surgery
Brief Title: Comparing the Establishment of Operation Space Between High Position and Low Position in Endoscopic Thyroid Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Bo Wang,MD, Clinical Professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Space H and L
Record Dates: First submitted 2018-06-24; First posted 2018-07-05 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Thyroid Cancer; Endoscopy
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high position space group (Experimental): The left and right Trocar meet at the level of the sternum angle and begin to establish the operating space.
  Interventions: Procedure: high position space group
- low position space group (Experimental): The left and right Trocar meet under the sternum angle and begin to establish the operating space.
  Interventions: Procedure: low position space group

INTERVENTIONS:
Procedure: high position space group — The left and right Trocar meet at the level of the sternum angle and begin to establish the operating space.
  Arms: high position space group
Procedure: low position space group — The left and right Trocar meet under the sternum angle and begin to establish the operating space.
  Arms: low position space group

SUMMARY:
Patients in our department endoscopic thyroidectomy were randomly divided into high position and low position established operating space group established operating space group. The thyroid size, patient BMI, operation time, and intraoperative blood loss were compared between the two groups.

DETAILED DESCRIPTION:
Patients in our department endoscopic thyroidectomy were randomly divided into high position and low position established operating space group established operating space group.The sternum angle level is used as the dividing line between the two groups。The thyroid size, patient BMI, operation time, and intraoperative blood loss were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with endoscopic thyroid surgery
* No previous neck surgery

Exclusion Criteria:

* Patients undergoing lateral neck lymph node dissection during the same period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
Intercostal arterial bleeding | During surgery
  The number of intercostal artery bleeding
Thyroidectomy time | During surgery
  Time to complete removal of thyroid gland specimens starting from the establishment of the operating space (minutes)

SECONDARY OUTCOMES:
Thyroid volume | Before surgery
  Thyroid volume calculated by preoperative ultrasound
Patient's BMI | Before surgery
  BMI equals body weight divided by height squared
Assessment of skin sensory abnormalities | two months after surgery
  According to the visual scoring method, it was divided into 1-10 points and evaluated by the patient two months after surgery. The score of 10 points was the same as before surgery, and 0 points showed serious discomfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China